CLINICAL TRIAL: NCT07058545
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of CJC-1134-PC Injection Administered Once Weekly in Antidiabetic Treatment-naive Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: A Study of CJC-1134-PC Injection in Antidiabetic Treatment-naive Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changshan ConjuChem BioPharmaceutical Research and Development (Hebei) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSCJC DM302
Record Dates: First submitted 2025-06-18; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus - Poor Control

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CJC-1134-PC (Experimental): Injection, 0.2ml/2mg (prefilled pen)
  Interventions: Drug: CJC-1134-PC Injection
- Placebo (Placebo Comparator): Injection, 0.2ml/0mg (prefilled pen)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CJC-1134-PC Injection — Double-blind Treatment Period: 0.2ml (2mg) once weekly ×24 weeks (Week 1 to Week 24); Open-label Treatment Period: 0.2ml (2mg) once weekly ×28 weeks (Week 25 to Week 52)
  Arms: CJC-1134-PC
Drug: Placebo — Double-blind Treatment Period: 0.2ml (0mg) once weekly ×24 weeks (Week 1 to Week 24); Open-label Treatment Period: 0.2ml (2mg) once weekly ×28 weeks (Week 25 to Week 52)
  Arms: Placebo

SUMMARY:
This study is a Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of CJC-1134-PC Injection Administered Once Weekly in Antidiabetic Treatment-naive Patients with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for the study only if all the following inclusion criteria were met:

1. Males or females aged 18 - 70 years (inclusive) at screening;
2. Subjects with body mass index (BMI) ≥ 20 kg/ m2 and ≤ 40 kg/ m2.
3. Subjects diagnosed with type 2 diabetes mellitus according to 1999 World Health Organization (WHO) criteria;
4. Subjects who had not received anti-diabetic therapy (including oral and injectable drugs, Chinese herbs for hypoglycemic purposes, and investigational anti-diabetic products, etc.) within 3 months prior to screening and had used anti-diabetic drugs for no more than 2 weeks since diagnosis;
5. Subjects with a stable lifestyle prior to screening, e.g. no significant changes in diets and physical exercise;
6. Subjects with fasting plasma glucose (FPG) or fasting serum glucose ≤13.9 mmol/L (250 mg/dL) at screening as determined by the local laboratory (study center) and FPG≤13.9 mmol/L (250 mg/dL) as determined by the central laboratory;
7. Subjects with HbA1c levels ≥ 7.0% and ≤ 11.0% at screening as determined by the local laboratory (study center), and HbA1C ≥ 7.0% and ≤ 11.0% as determined by the central laboratory;
8. Patients who were able to understand the procedures and methods of the study, willing to strictly comply with the clinical trial protocol, and voluntarily signed an informed consent form (ICF).

Exclusion Criteria:

Subjects were not eligible for the study if they met any of the following criteria:

Prior and concomitant diseases

1. Diagnosed as type 1 diabetes mellitus, diabetes mellitus due to pancreatic injury, or secondary diabetes mellitus caused by other diseases (e.g., acromegaly or Cushing syndrome);
2. History of acute and chronic pancreatitis prior to screening or current history of acute and chronic pancreatitis;
3. Presence of active gallbladder or biliary tract disease within 1 year prior to screening (active means presence of relevant symptoms);
4. Family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (family refers to first-degree blood relatives);
5. Presence of malignant tumors in the past 5 years (except for cured skin basal cell carcinoma and carcinoma in situ of cervix).
6. Decompensated cardiac insufficiency (New York Heart Association class III or IV) either within the 6 months prior to screening or currently;
7. History of myocardial infarction, coronary artery bypass grafting, coronary stenting, haemorrhagic or ischaemic stroke (except lacunar cerebral infarction), or hospitalisation for unstable angina pectoris or transient ischaemic attack within 6 months prior to screening;
8. Uncontrolled and severe arrhythmia [e.g., degree II or III AV block, prolonged QT interval (QTc > 450 ms)] within 6 months prior to screening and judged by the investigator to be unsuitable for participation in this trial;
9. Severe diabetic neuropathy within 6 months prior to screening;
10. Proliferative diabetic retinopathy diagnosed within 6 months before or at the time of screening, either confirmed by non-mydriatic fundus photography or by pharmacologically dilated fundus examination performed by an ophthalmic healthcare provider (unless contraindicated), or with a history of laser treatment for proliferative diabetic retinopathy within the 6 months prior to screening;
11. Diabetic ketoacidosis or hyperglycemic hyperosmolar state occurring within 6 months prior to screening and up to randomization;
12. Previous major gastric-related surgery (e.g., major or total gastrectomy, sleeve gastrectomy, gastric bypass), current history of significant gastrointestinal conditions (such as active ulcers, gastroparesis, pyloric obstruction, intestinal obstruction, inflammatory bowel disease, etc.), or chronic gastrointestinal diseases requiring prolonged use of medications that directly affect gastrointestinal motility and are deemed unsuitable for participation in this trial by the investigator;
13. Severe trauma or major surgery occurring within 1 month prior to screening up to randomization, or the systemic use of antimicrobial agents, as determined by the investigator, which may potentially impact blood glucose control; Prohibited therapies and/or drugs
14. Subjects who were using weight-loss drugs, and those with significant changes (at least 10%) in body weight 3 months prior to screening;
15. Subjects who received treatment with any other investigational drug or device within 3 months prior to screening;
16. Subjects who received treatment with systemic glucocorticoids (other than inhaled or topical glucocorticoids) or growth hormone within 3 months prior to screening;
17. Subjects who were using warfarin at the time of screening and were unable to discontinue it for the duration of the study; Laboratory results
18. Systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg after 5 minutes of sedentary rest at the time of screening or on the day of randomization [if the above criteria were not met, the test could be repeated twice (each time more than 1 minute apart), and the average of the three tests could be used to assess against the aforementioned criteria again];
19. Estimated glomerular filtration rate (eGFR) < 60 mL/min (see Appendix 14.2 of the Clinical Study Protocol [V1.2/15Dec2020] for the formula) or urinary protein qualitative assessment ≥++;
20. Subjects with alanine aminotransferase (ALT) or/and aspartate aminotransferase (AST) > 2.5 × ULN (upper limit of normal), or total bilirubin level > 1.5 × ULN;
21. Subjects currently presenting with uncontrolled thyroid dysfunction despite a stable medication dosage (defined as a stable dose for 4 weeks or more) or clinically significant abnormalities in thyroid function test results (thyroid-stimulating hormone [TSH], serum free thyroxine [FT4], and free triiodothyronine [FT3]) at the time of screening;
22. Subjects currently suffering from anaemia (haemoglobin <120 g/L for men and <110 g/L for women) or other conditions that affected HbA1c testing;
23. Subjects with fasting triglyceride < 5.64 mmol/L (<500 mg/dL);
24. Serum amylase or lipase >3×ULN;
25. Subjects who were positive for Hepatitis B surface antigen, Hepatitis C antibody and human immunodeficiency virus (HIV) antibody (weakly positive was considered positive); Gender and reproductive status
26. Subjects with positive pregnancy test;
27. Subjects who were pregnant or lactating at enrollment;
28. Female subjects of childbearing potential or male subjects with sexual partners of childbearing potential, who were unwilling to take medically recognized effective contraceptive measures (including condoms with spermicide, vaginal diaphragm, oral or injectable contraceptives) during the study and within 3 months after discontinuation; Other criteria
29. Alcoholics [>2 units of alcohol per day and >14 units per week (1 unit of alcohol is equivalent to 150 mL of wine, 350 mL of beer, or 50 mL of spirits)] or individuals with a history of drug abuse;
30. Subjects with blood donation or transfusion ≥ 400 mL within 3 months before screening;
31. Subjects with mental deficiency or serious mental illness which might affect the signing of informed consent form and the compliance with the study protocol;
32. Subjects who refused to take anti-diabetic drugs only specified in the protocol throughout the study;
33. Hypersensitivity to Albenatide, human albumin (API for Albenatide formulations), Amaryl® (glimepiride tablets) or related excipients;
34. Intolerance to Albenatide or Amaryl® (glimepiride tablets);
35. Other conditions that are deemed inappropriate by the investigator to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at the end of double-blind treatment period. | Week 25 visit
  The double-blind treatment period ended at the 25-week visit.

SECONDARY OUTCOMES:
Proportion of subjects with HbA1c <7.0% at the end of the double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Proportion of subjects with HbA1c <6.5% at the end of the double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting weight at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting waist circumference at the end of double-blind /open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting plasma glucose at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting proinsulin at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting insulin at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting C-peptide at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (total cholesterol) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (low-density lipoprotein [LDL]) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (high-density lipoprotein [HDL]) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (triglycerides) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in fasting lipids (LDL/HDL ratio) at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in systolic blood pressure [SBP] at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in diastolic blood pressure [DBP] at the end of double-blind treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in 6-point finger-stick blood glucose at the end of double-blind/open-label treatment period. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in blood AST at the end of double-blind/open-label treatment period in patients diagnosed with fatty liver on screening imaging. | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Changes from baseline in blood ALT at the end of double-blind/open-label treatment period in patients diagnosed with fatty liver on screening imaging | Week 25 visit, and week 53 visit.
  The double-blind treatment period ended at the 25-week visit, and the open-label treatment period ended at the 53-week visit.
Change from baseline in HbA1c at the end of open-label treatment period. | Week 53 visit.
  The open-label treatment period ended at the 53-week visit.

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Prof., Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No